CLINICAL TRIAL: NCT00695279
Title: Long Term Follow Up Of Patients Who Have Received Gene Therapy Or Gene Marked Products at St. Jude Children's Research Hospital
Brief Title: Long Term Follow Up Of Patients Who Have Received Gene Therapy Or Gene Marked Products
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GENEFU; NCI-2021-10844 (Registry Identifier: NCI)
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Severe Combined Immunodeficiency; Malignancy, Hematologic; Neuroblastoma; Neoplasm; Mucopolysaccharidosis I
Keywords: Gene therapy
MeSH Terms: conditions — Severe Combined Immunodeficiency; Hematologic Neoplasms; Neuroblastoma; Neoplasms; Mucopolysaccharidosis I | interventions — Phlebotomy; Follow-Up Studies; Prospective Studies; Cancer Vaccines; Biological Specimen Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Venipuncture
  Interventions: Procedure: Venipuncture

INTERVENTIONS:
Procedure: Venipuncture — Blood draw
  Other Names: Follow-Up Studies; Prospective Studies; Cancer vaccines; Biological Specimen Banks

SUMMARY:
This protocol (GENEFU) provides a mechanism for the 15-year followup period that the FDA requires for all participants in gene transfer protocols and assures that adequate followup can be maintained for a wide variety of participants on different individual gene therapy protocols at St. Jude Children's Research Hospital.

GENEFU serves as an umbrella protocol for long-term follow-up (LTFU) for recipients of gene therapy/gene marked (GT/GM) products at St. Jude Children's Research Hospital. The FDA has recommended methods to assess the risk of delayed adverse events after GT/GM and has provided specific requirements regarding the duration and design of LTFU observations. This protocol is intended to provide LTFU in accordance with the FDA guidelines for those who received a GT/GM product as part of a St. Jude-sponsored clinical trial or compassionate use treatment plan. The protocol calls for a physical examination or general health evaluation and collection of required blood samples annually for up to 15 years after the last receipt of a GT/GM product.

Goals will be to obtain clinical histories in order to detect late clinical outcomes suggestive of retroviral or lentiviral disease, including but not limited to cancer/second malignancies, neurologic disorders, autoimmune disorders, and hematologic disorders. Blood samples will be archived and tested when clinically or scientifically indicated, as in the event of development of a second malignancy. This prospective cohort study will utilize descriptive statistics in the analysis of long-term late effects outcomes. It offers a uniform approach to long-term safety monitoring in research participants who have received a gene-transduced product as part of St. Jude-sponsored GT or GM protocols and compassionate use treatment plans.

DETAILED DESCRIPTION:
Secondary objectives include the following: to obtain and archive blood samples to 1) detect frequency of vector marking in peripheral blood mononuclear cells when clinically or scientifically indicated, such as in the event of participant development of second malignancy, autoimmune disease, hematologic abnormality, or neurologic event, and; 2) To obtain and archive blood samples to detect and characterize clonal proliferation events occurring in gene transfer trials when clinically or scientifically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Has received an integrating retroviral or lentiviral vector based GT/GM product at St. Jude Children's Research Hospital within the past 15 year time period. Patient is no later than 15 years post receipt of GT/GM product.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gene therapy recipient patients
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-01-04 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Obtain histories for detection of significant delayed medical events in research participants who have received an integrating vector-based gene therapy/gene marked product at St. Jude Children's Research Hospital (SJCRH). | 30 years
  Obtain histories for detection of significant delayed medical events including hematologic, malignant, autoimmune, and neurologic events in research participants who have received an integrating vector-based gene therapy/gene marked product at St. Jude Children's Research Hospital (SJCRH).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gottschalk, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols